CLINICAL TRIAL: NCT06236503
Title: Effect of Daily Transcranial Direct Current Stimulation on the Cognitive Evolution of Patients in an Altered State of Consciousness
Brief Title: Effect of Transcranial Direct Current Stimulation in Altered States of Consciousness
Acronym: tDCS-GCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Viviana Lo Buono, Dr., IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: tDCS-GCA
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Neurologic Disorder; Brain Injuries
MeSH Terms: conditions — Nervous System Diseases; Brain Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real Stimulation (Experimental): Time A. Behavioral assessment using the Coma Recovery Scale-R (CRS-R). Time B. Transcranial Direct Current Stimulation (tDCS). Frontal stimulation for 20 minutes with the anode placed on the international electrode 10-20 position and the cathode on the right supraorbital region. Stimulation will be repeated once a day, 5 days a week, for 4 weeks. Time C. Behavioral assessment using the coma recovery scale-R (CRS-R). Rest Period 2 months.
  Interventions: Behavioral: Real Stimulation
- Placebo Stimulation (Placebo Comparator): Time A. Behavioral assessment using the Coma Recovery Scale-R (CRS-R). Time B. Transcranial Direct Current Stimulation (tDCS). Frontal stimulation for 5 seconds with the anode placed on the international electrode position and the cathode on the right supraorbital region. Stimulation will be repeated once a day, 5 days a week, for 4 weeks. · Time C: Behavioral assessment using the Coma Recovery Scale-R (CRS-R). Time D: Behavioral assessment using the coma Recovery Scale-R (CRS-R).
  Interventions: Behavioral: Placebo Stimulation

INTERVENTIONS:
Behavioral: Real Stimulation — Time A: Behavioral assessment using the Coma Recovery Scale-R (CRS-R). · Time B:
  Transcranial Direct Current Stimulation (tDCS). Frontal stimulation for 20 minutes with the anode placed on the international electrode position and the cathode on the right supraorbital region. Stimulation will be repeated once a day, 5 days a week, for 4 weeks. · Time C. Behavioral assessment using the Coma Recovery Scale-R (CRS-R). Rest Period: 2 months.
  Arms: Real Stimulation
Behavioral: Placebo Stimulation — Time A: Behavioral assessment using the Coma Recovery Scale-R (CRS-R). Time B. Transcranial Direct Current Stimulation (tDCS). Frontal stimulation for 5 seconds with the anode placed on the electrode 10-20 position and the cathode on the right supraorbital region. Stimulation will be repeated once a day, 5 days a week, for 4 weeks. · Time C. Behavioral assessment using the Coma recovery Scale-R (CRS-R). Time D. Behavioral assessment using the Coma Recovery Scale-R (CRS-R).
  Arms: Placebo Stimulation

SUMMARY:
Transcranial Direct Current Stimulation (tDCS) is a non-invasive, painless brain stimulation treatment that uses low-intensity direct electrical currents to stimulate specific parts of the brain. Transcranial Direct Current Stimulation (tDCS) can both facilitate anodic stimulation and inhibit cathodic stimulation specific brain areas since many neurological and psychiatric disorders are connected to hypoactivity or hyperactivity in specific areas of the nervous system. This phenomenon is based on two processes: the reorganization of functional neural circuits and their reconstruction. In light of the studies mentioned above, it is presumed that Transcranial Direct Current Stimulation (tDCS) can be a valuable tool to facilitate the process of neuroplasticity in individuals with chronic neurological diseases and in patients with impaired consciousness following severe brain injury. A previous study demonstrated that a single session of transcranial direct current electrical stimulation could temporarily improve signs of consciousness in patients in a minimally conscious state (MCS)

DETAILED DESCRIPTION:
Transcranial Direct Current Stimulation (tDCS) is a non-invasive, painless brain stimulation treatment that uses low-intensity direct electrical currents to stimulate specific parts of the brain. Transcranial Direct Current Stimulation (tDCS) can both facilitate anodic stimulation and inhibit cathodic stimulation specific brain areas since many neurological and psychiatric disorders are connected to hypoactivity or hyperactivity in specific areas of the nervous system. This phenomenon is based on two processes: the reorganization of functional neural circuits and their reconstruction. In light of the studies mentioned above, it is presumed that Transcranial Direct Current Stimulation can be a valuable tool to facilitate the process of neuroplasticity in individuals with chronic neurological diseases and in patients with impaired consciousness following severe brain injury. A previous study demonstrated that a single session of transcranial direct current electrical stimulation could temporarily improve signs of consciousness in patients in a minimally conscious state (MCS).

The application of weak currents can interact with neural processing, modify plasticity and entrain brain networks, and that this in turn can modify behaviour. The technique is now widely employed in basic and translational research, and increasingly is also used privately in sport, the military and recreation. The proposed capacity to augment recovery of brain function, by promoting learning and facilitating plasticity, has motivated a burgeoning number of clinical trials in a wide range of disorders of the nervous system. In this experimental study, cortical brain areas will be stimulated using transcranial direct current stimulation (tDCS) in patients with impaired consciousness following severe brain injury.

The main aim of this study is to determine whether the long-term effects of Transcranial Direct Current Stimulation (tDCS) stimulation can persist over time and whether this technique could be applied in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a minimally conscious state will be evaluated and stimulated, provided that written informed consent is obtained from a family member.

Exclusion Criteria:

patients in coma patients with metallic brain implants, craniotomy or pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale-R (CRS-R). | 4 weeks
  Behavioral assessment using the Coma Recovery Scale-R (CRS-R) for for the assessment of changes in the state of consciousness

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italia, Italy

IPD SHARING:
Plan to Share IPD: No